CLINICAL TRIAL: NCT02923349
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of INCAGN01949 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety Study of INCAGN01949 in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 1949-101; 2016-002079-93 (EudraCT Number)
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignancies; Metastatic Cancer
Keywords: Solid tumor; adenocarcinoma of the endometrium; ovarian cancer; renal cell carcinoma; melanoma; non-small cell lung cancer; OX40; immunoglobulin G monoclonal antibody
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCAGN01949 (Experimental)
  Interventions: Drug: INCAGN01949

INTERVENTIONS:
Drug: INCAGN01949 — Initial cohort dose of INCAGN01949 monotherapy at the protocol-defined starting dose, with subsequent cohort escalations based on protocol-specific criteria. The recommended dose will be taken forward into expansion cohorts.

SUMMARY:
The purpose of this study is to determine the safety and tolerability and assess preliminary efficacy of INCAGN01949 in subjects with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Subjects who have disease progression after treatment with available therapies that are known to confer clinical benefit, or who are intolerant to treatment, or who refuse standard treatment. There is no limit to the number of prior treatment regimens.
* Part 1: Subjects with advanced or metastatic solid tumors.
* Part 2: Subjects with advanced or metastatic adenocarcinoma of the endometrium, ovarian cancer, renal cell carcinoma, melanoma, and non-small cell lung cancer.
* Presence of measureable disease based on RECIST v1.1.
* Eastern Cooperative Oncology Group performance status 0 or 1.

Exclusion Criteria:

* Laboratory and medical history parameters not within the protocol-defined range.
* Receipt of anticancer medications or investigational drugs within the protocol-defined intervals before the first administration of study drug.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior immunotherapy) and/or complications from prior surgical intervention before starting therapy.
* Receipt of a live vaccine within 30 days of planned start of study drug.
* Active autoimmune disease that required systemic treatment in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Janik, MD, Study Director — Incyte Corporation
Locations (8):
- United States (4):
  - Rutgers, The State University of New Jersey, New Brunswick, New Jersey
  - New York University Clinical Cancer Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Spain
- University Hospital of Laussane (CHUV), Lausanne, Switzerland
- United Kingdom (2):
  - University College Hospital, London
  - University of Oxford, Oxford

REFERENCES:
- [Derived] Davis EJ, Martin-Liberal J, Kristeleit R, Cho DC, Blagden SP, Berthold D, Cardin DB, Vieito M, Miller RE, Hari Dass P, Orcurto A, Spencer K, Janik JE, Clark J, Condamine T, Pulini J, Chen X, Mehnert JM. First-in-human phase I/II, open-label study of the anti-OX40 agonist INCAGN01949 in patients with advanced solid tumors. J Immunother Cancer. 2022 Oct;10(10):e004235. doi: 10.1136/jitc-2021-004235. PMID 36316061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 different sites in US, 1 site in Switzerland,1 site in Spain and 2 sites in the United Kingdom.
Pre-assignment Details: A total of 129 participants were screened for this study, of which 42 participants were screen failures and 87 participants were randomized to treatment.
Groups:
- PART 1 Dose 1 (7 mg): INCAGN01949 7mg administered intravenously over a 30-minute period on Day 1 of each cycle in subjects with advanced or metastatic solid tumors
- PART 1 Dose 2 (20 mg): INCAGN01949 20mg administered intravenously over a 30-minute period on Day 1 of each cycle in subjects with advanced or metastatic solid tumors
- PART 1 Dose 3 (70 mg): INCAGN01949 70mg administered intravenously over a 30-minute period on Day 1 of each cycle in subjects with advanced or metastatic solid tumors
- PART 1 Dose 4 (200 mg): INCAGN01949 200mg administered intravenously over a 30-minute period on Day 1 of each cycle in subjects with advanced or metastatic solid tumors
- PART 1 Dose 5 (350 mg): INCAGN01949 350mg administered intravenously over a 30-minute period on Day 1 of each cycle in subjects with advanced or metastatic solid tumors
- PART 1 Dose 6 (700 mg): INCAGN01949 700mg administered intravenously over a 30-minute period on Day 1 of each cycle in subjects with advanced or metastatic solid tumors
- PART 1 Dose 7 (1400 mg): INCAGN01949 1400mg administered intravenously over a 30-minute period on Day 1 of each cycle in subjects with advanced or metastatic solid tumors
Period: Overall Study
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Started | 4 | 4 | 22 | 18 | 23 | 12 | 4
Completed | 0 | 0 | 5 | 2 | 4 | 5 | 1
Not Completed | 4 | 4 | 17 | 16 | 19 | 7 | 3
Not completed — Other | 1 | 2 | 4 | 1 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 8 | 10 | 12 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 2 | 4 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg) | Total
Number analyzed (Participants) | 4 | 4 | 22 | 18 | 23 | 12 | 4 | 87
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 54.3 (16.24) | 63.8 (12.63) | 56.8 (14.27) | 58.9 (12.78) | 58.1 (12.44) | 61.3 (9.93) | 52.8 (24.50) | 58.2 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 14 | 12 | 17 | 3 | 2 | 53
  Male | 2 | 1 | 8 | 6 | 6 | 9 | 2 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 4 | 3 | 19 | 17 | 23 | 9 | 4 | 79
  Asian | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 4
  Other | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Black/African American | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 4 | 4 | 19 | 16 | 22 | 11 | 2 | 78
  Not Reported | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Maximum Observed Concentration (Cmax) of INCAGN01949 in Plasma
Description: To evaluate the Cmax of INCAGN01949 in subjects with advanced or metastatic solid tumors.
Time Frame: Pre-infusion for cycles 1,2,3,4,5,6 and 7, 10-minutes, 4 hrs, 24 hrs post-infusion, Day 8 for cycles 1 & 6
Population: The PK evaluable population will include all subjects who received at least 1 dose of INCAGN01949 and provided at least 1 post dose sample (1 PK measurement).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 4 | 4 | 21 | 17 | 21 | 7 | 4
ng/ml | 1630 (735) | 5820 (324) | 22300 (32800) | 39200 (10300) | 84900 (76700) | 207000 (45500) | 347000 (130000)

2. Secondary Outcome: Area Under the Single-dose Concentration-time Curve (AUC0-t) of INCAGN01949
Description: To evaluate the AUC0-t of INCAGN01949 in subjects with advanced or metastatic solid tumors
Time Frame: Pre-infusion for cycles 1,2,3,4,5,6 and 7, 10-minutes, 4 hrs, 24 hrs post-infusion, Day 8 for cycles 1 & 6
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 4 | 4 | 21 | 17 | 21 | 7 | 4
ug*hr/mL
  cycle 1 | 185 (81.7) | 904 (197) | 2370 (841) | 5400 (1820) | 10000 (5600) | 28300 (7720) | 61600 (9130)
  cycle 6: number analyzed (Participants) | 2 | 0 | 4 | 3 | 0 | 0 | 0
  cycle 6 | 427 (9.21) |  | 5490 (1560) | 10700 (6560) |  |  |

3. Secondary Outcome: Objective Response Rate Per RECIST and Modified RECIST
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) per RECIST v1.1 and mRECIST v1.1. by investigator determination.
Time Frame: Baseline and every 8 weeks,up to 11 months
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCAGN01949.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 4 | 4 | 22 | 18 | 23 | 12 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Duration of Response Per RECIST and Modified RECIST
Description: as for outcome 3
Time Frame: Baseline and every 8 weeks, up to 11 months
Population: The Full Analysis Set population included all subjects enrolled in the study who received at least 1 dose of INCAGN01949. Median was not estimable due to insufficient number of participants with response
Measure: Median (Full Range); unit: days
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0
days |  |  |  |  |  | 192 (192) [192 to 192] |

5. Secondary Outcome: Progression-free Survival Per RECIST and Modified RECIST
Description: as for outcome 3
Time Frame: Baseline and every 8 weeks, up to 11 months
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCAGN01949.
Measure: Median (Full Range); unit: Days
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 4 | 4 | 22 | 18 | 23 | 12 | 4
Days | 57 (55) [55 to 59] | 47.5 (29) [29 to 112] | 54.0 (23) [23 to 216] | 56.0 (26) [26 to 281] | 52.0 (1) [1 to 166] | 125.0 (21) [21 to 298] | 46.5 (42) [42 to 53]

6. Secondary Outcome: Duration of Disease Control Per RECIST and Modified RECIST
Description: as for outcome 3
Time Frame: Baseline and every 8 weeks, up to 11 months
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCAGN01949. Median was not estimable due to insufficient number of participants with CR, PR, and SD
Measure: Median (Full Range); unit: Days
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 1 | 1 | 8 | 7 | 3 | 7 | 0
Days | 0 [0 to 0] | 57 [57 to 57] | 64 [1 to 160] | 57 [1 to 225] | NA [1 to 112] — The numbers reported were censored durations of stable disease for the participants. Median is not estimable as Kaplan-Meier method requires at least 1 event to determine where the curve hits 50% rate of estimated durations | 120 [1 to 249] |

7. Primary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment
Time Frame: From screening through 60 days after end of treatment, up to 11 months
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCAGN01949.
Measure: Count of Participants; unit: Participants
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 4 | 4 | 22 | 18 | 23 | 12 | 4
Participants | 4 | 4 | 21 | 17 | 22 | 11 | 4

8. Secondary Outcome: Time to Maximum Concentration of INCAGN01949 in Plasma
Description: To evaluate the Tmax of INCAGN01949 in subjects with advanced or metastatic solid tumors.
Time Frame: Pre-infusion for cycles 1,2,3,4,5,6 and 7, 10-minutes, 4 hrs, 24 hrs post-infusion, Day 8 for cycles 1 & 6
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 4 | 4 | 21 | 17 | 21 | 7 | 4
hr
  cycle 1 | 0.64 [0.6 to 4.4] | 2.53 [0.55 to 4.5] | 4.3 [0.50 to 25.2] | 0.63 [0.5 to 4.5] | 0.6 [0.0 to 194] | 0.7 [0.53 to 4.2] | 0.73 [0.0 to 2.43]
  cycle 6: number analyzed (Participants) | 2 | 0 | 4 | 3 | 0 | 0 | 0
  cycle 6 | 0.78 [0.75 to 0.8] |  | 0.63 [0.50 to 4.3] | 0.61 [0.55 to 4.8] |  |  |

9. Secondary Outcome: Summary of Trough Concentrations(Cmin) of INCAGN01949
Description: To evaluate the Cmin of INCAGN01949 in subjects with advanced or metastatic solid tumors. Cmin is the minimum observed concentration of INCAGN1949
Time Frame: Pre-infusion for cycles 1,2,3,4,5,6 and 7, 10-minutes, 4 hrs, 24 hrs post-infusion, Day 8 for cycles 1 & 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
Number analyzed (Participants) | 4 | 4 | 22 | 18 | 23 | 12 | 4
ng/mL
  cycle 2: number analyzed (Participants) | 4 | 4 | 20 | 17 | 18 | 7 | 3
  cycle 2 | 303 (202) | 1890 (1570) | 3620 (1550) | 8880 (4510) | 17000 (8040) | 41000 (13000) | 117000 (19300)
  cycle 3: number analyzed (Participants) | 3 | 3 | 17 | 14 | 15 | 4 | 4
  cycle 3 | 753 (163) | 1520 (225) | 5620 (3280) | 14300 (7740) | 29400 (18400) | 77800 (27900) | 163000 (32900)
  cycle 4: number analyzed (Participants) | 3 | 2 | 12 | 12 | 8 | 3 | 2
  cycle 4 | 895 (80.2) | 1780 (318) | 5110 (2850) | 17900 (13200) | 42200 (28500) | 84600 (17700) | 282000 (165000)
  cycle 6: number analyzed (Participants) | 2 | 0 | 4 | 4 | 3 | 0 | 0
  cycle 6 | 785 (39.6) |  | 9150 (2420) | 19600 (13100) | 43400 (26500) |  |
  cycle 7: number analyzed (Participants) | 0 | 0 | 2 | 4 | 0 | 0 | 0
  cycle 7 |  |  | 10200 (2190) | 21600 (10600) |  |  |

ADVERSE EVENTS:
Time Frame: From screening through 60 days after end of treatment, up to 11 months
Arm/Group | PART 1 Dose 1 (7 mg) | PART 1 Dose 2 (20 mg) | PART 1 Dose 3 (70 mg) | PART 1 Dose 4 (200 mg) | PART 1 Dose 5 (350 mg) | PART 1 Dose 6 (700 mg) | PART 1 Dose 7 (1400 mg)
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/4 | 2/22 | 4/18 | 2/23 | 3/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4 | 8/22 | 9/18 | 9/23 | 5/12 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 21/22 | 17/18 | 22/23 | 10/12 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PART 1 Dose 1 (7 mg) (N=4) | PART 1 Dose 2 (20 mg) (N=4) | PART 1 Dose 3 (70 mg) (N=22) | PART 1 Dose 4 (200 mg) (N=18) | PART 1 Dose 5 (350 mg) (N=23) | PART 1 Dose 6 (700 mg) (N=12) | PART 1 Dose 7 (1400 mg) (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 2 | 3 | 0
Myelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PART 1 Dose 1 (7 mg) (N=4) | PART 1 Dose 2 (20 mg) (N=4) | PART 1 Dose 3 (70 mg) (N=22) | PART 1 Dose 4 (200 mg) (N=18) | PART 1 Dose 5 (350 mg) (N=23) | PART 1 Dose 6 (700 mg) (N=12) | PART 1 Dose 7 (1400 mg) (N=4)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 4 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2 | 1 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 1 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2 | 5 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 4 | 6 | 4 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 5 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 6 | 4 | 7 | 3 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 4 | 3 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 3 | 3 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 2
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 6 | 7 | 8 | 4 | 2
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 (5) | 3 | 6 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 3 | 0 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 2 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0 | 2 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 5 | 3 | 4 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 0 | 2 | 2 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02923349/Prot_001.pdf
  • Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT02923349/SAP_000.pdf